CLINICAL TRIAL: NCT03593408
Title: Pharmacokinetics of Sedatives and Analgesics During Extracorporeal Membrane Oxygenation (ECMO) Support
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Viviane Nasr, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00028380
Record Dates: First submitted 2018-06-26; First posted 2018-07-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Drug Effect
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Midazolam; Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients on ECMO Support
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl; Drug: Midazolam; Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine — Administered for sedation management per hospital protocol
Drug: Fentanyl — Administered for sedation management per hospital protocol
Drug: Midazolam — Administered for sedation management per hospital protocol
Drug: Morphine — Administered for sedation management per hospital protocol

SUMMARY:
This study will measure plasma concentrations of dexmedetomidine, fentanyl, morphine and midazolam in pediatric patients supported with extracorporeal membrane oxygenation (ECMO) aiming to understand the pharmacokinetics of these drugs in this setting.

ELIGIBILITY:
Inclusion Criteria:

* supported on ECMO
* receiving one or a combination of the following drugs dexmedetomidine, fentanyl, midazolam or morphine as part of sedation management

Exclusion Criteria:

-none

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients who present to Boston Children's Hospital (BCH) and supported on ECMO and receiving one or a combination of the following drugs dexmedetomidine, fentanyl, midazolam or morphine as part of the sedation management.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma concentrations of dexmedetomidine | Throughout the duration of sedation management with dexmedetomidine at baseline, 30, 60, 120 minutes and then at 4, 6, 12 hours after each bolus or change in infusion and then at 30,60, 90, 120, 240minutes and 4 hours after the drug is stopped
change in plasma concentrations of fentanyl | Throughout the duration of sedation management with fentanyl at baseline, 30, 60, 120 minutes and then at 4, 6, 12 hours after each bolus or change in infusion and then at 30,60, 90, 120, 240minutes and 4 hours after the drug is stopped
change in plasma concentrations of morphine | Throughout the duration of sedation management with morphine at baseline, 30, 60, 120 minutes and then at 4, 6, 12 hours after each bolus or change in infusion and then at 30,60, 90, 120, 240minutes and 4 hours after the drug is stopped
change in plasma concentrations of midazolam | Throughout the duration of sedation management with midazolam at baseline, 30, 60, 120 minutes and then at 4, 6, 12 hours after each bolus or change in infusion and then at 30,60, 90, 120, 240minutes and 4 hours after the drug is stopped

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Nasr, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States